CLINICAL TRIAL: NCT01795248
Title: The Impact of Liraglutide on Glucose Tolerance and the Risk of Type 2 Diabetes in Women With Previous Gestational Diabetes Mellitus
Brief Title: The Impact of Liraglutide on Glucose Tolerance and the Risk of Type 2 Diabetes in Women With Previous Pregnancy-induced Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tina Vilsboll (Other)
Collaborators: Novo Nordisk A/S (Industry); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Herlev Hospital (Other); Hillerod Hospital, Denmark (Other); University of Copenhagen (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Tina Vilsboll, Dr. Tina Vilsbøll, DMSc, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GDM-TREAT; 2012-001371-37 (EudraCT Number)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; incretin; glucose homeostasis; GLP-1; type 2 diabetes mellitus; liraglutide; Victoza
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide (Experimental): 1.8 mg liraglutide, subcutaneous, once-daily for five years
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo, subcutaneous, once-daily for one year
  Interventions: Drug: Placebo
- Control (No Intervention): Control without previous GDM.

INTERVENTIONS:
Drug: Liraglutide — 1.8 mg liraglutide
  Other Names: Victoza; NN2211
  Arms: Liraglutide
Drug: Placebo — Liraglutide without the GLP-1 analogue
  Arms: Placebo

SUMMARY:
It is well-known that women with previous gestational diabetes mellitus are in risk of developing type 2 diabetes later in life; approximately half of the women develop overt type 2 diabetes within the first 10 years after pregnancy. Knowing this, we want to examine the effect of the type 2 diabetes medicine, liraglutide (Victoza), in women with previous gestational diabetes with the aim of reducing the risk of developing type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria for women with previous GDM:

* Informed oral and written consent
* Previous diagnosis of GDM according to current Danish guidelines (mainly PG concentrationa t 120 min after 75 g OGTT ≥ 9.0 mM) during pregnancy within the last 5 years
* Age >18 years
* 25 kg/m2 < BMI < 45 kg/m2
* NGT, IFG and or IGT
* Safe contraception and negative pregnancy test

Exclusion Criteria for women with previous GDM:

* Patients with diabetes
* HbA1c ≥6.5%
* Patients with previous pancreatitis or previous neoplasia
* Pregnant or breast feeding women
* Anaemia (haemoglobin <7 mM)
* Women planning to become pregnant within the next 5 years
* Women using other contraception than intrauterine device (IUD) or oral contraceptives. Women who do not use safe contraception will be offered application of an IUD.
* Women treated with statins, corticosteroids or other hormone therapy (except estrogens and gestagens)
* Ongoing abuse of alcohol or narcotics
* Impaired hepatic function (liver transaminases >3 times upper normal limit)
* Impaired renal function (se-creatinine >120 μM and/or albuminuria)
* Uncontrolled hypertension (systolic blood pressure >180 mmHg, diastolic blood pressure >100 mmHg)
* Any condition that the investigator feels would interfere with trial participation
* Receiving any investigational drug within the last 3 months

Inclusion criteria for women without previous GDM:

* Informed oral and written consent
* Age >18 years
* 25 kg/m2 < BMI < 45 kg/m2
* NGT
* Safe contraception and negative pregnancy test
* Pregnancy within the last ten years without GDM

Exclusion Criteria for women without previous GDM :

* Pregnant or breast feeding women
* Anaemia (haemoglobin <7 mM)

Inclusion Criteria for women without previous GDM and without NAFLD:

* Informed oral and written consent
* Age >18 years
* 25 kg/m2 < BMI < 45 kg/m2
* NGT
* At least one pregnancy witin the last ten years without GDM

Exclusion Criteria for women without previous GDM and without NAFLD:

* Pregnant or breast feeding women
* Anaemia (haemoglobin <7 mM)
* Steatosis as assessed by ultrasound scanning
* Recieving any investigational drug within the last 3 months
* Any condition that the investigator feels would interfere with the trial participation

Inclusion Criteria for women with biopsi-verified NAFLD:

* Informed oral and written consent
* Women with known NAFLD or NASH
* Age >18 years
* 25 kg/m2 < BMI < 45 kg/m2
* NGT
* At least one prior pregnancy

Exclusion Criteria for women with biopsi-verified NAFLD:

* women with established cirrhosis
* Pregnant or breast feedning women
* Anaemia (haemoglobin <7 mM)
* Women treated with statins, corticosteroids or other hormone therapy ( except oestrogens and gestagens)
* Ongoing abuse of alcohol or narcotics
* Impaired renal function (se-creatinine > 120 μM and/or albuminuria)
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg, diastolic blood presure > 100 mmHg)
* Any condition that the investigator feels would interfere with trial participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance | from baseline to 52 wks, 53 wks, 260 wks, and 261 wks
  Changes in glucose is measured by area under the curve for the plasma glucose excursion following a 4-hour 75 g oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Deterioration in glycaemic status | from baseline to 52 wks, 53, wks, 260 wks, and 261 wks
  Percentage of subjects in each treatment arm with normal glucose tolerance (NGT) at inclusion who develop impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) or type 2 diabetes; or with IFG or IGT who develop combined IFG/IGT; or with combined IFG/IGT who develop type 2 diabetes

OTHER OUTCOMES:
Changes in glycated hemoglobin | From baseline to 52 wks and 260 wks
  Changes in glycated hemoglobin (HbA1c). From normoglycaemic to prediabetic or type 2 diabetic and from prediabetic to type 2 diabetic or normoglycaemic.
Changes in anthropometric measurements | from baseline to 52 and 260 wks
  Changes in body mass index (BMI)(kg/m2), absolute body weight (kg), and waist:hip ratio
Changes in beta cell secretory responses | from baseline to 52, 53, 260, and 261 wks
  changes in area under the curve during OGTT and isoglycemic intravenous glucose infusion (IIGI), the homeostatic model assessment (HOMA) and pro-insulin ratio
Changes in insulin sensitivity | from baseline to 52, 53, 260, and 261 wks
  assessed by HOMA-IR and Matsuda insulin sensitivity index
Changes in incretin hormone secretion | baseline to 52, 53, 260, and 261 wks
  measured as fasting plasma concentrations and plasma responses of GLP-1, GLP2, and GIP and plasma glucagon during OGTT
Changes in incretin effect | baseline to 52, 53, 260, and 261 wks
  insulin and c-peptide responses after OGTT vs. IIGI
Changes in presence of non-alcoholic fatty liver disease (NAFLD) | baseline to 52 and 260 wks
  gamma-glutamyltranferase (GGT), intra-heptic fat, FGF-21, whole body and visceral fat mass/fat-free mass, circulating lipids, ultrasound scan and fibroscan
Changes in cardio-metabolic risk measures | baseline to 52 and 260 wks
  pro-collagen 3, GGT, Intra-hepatic fat, whole body and visceral fat mass/fat-free mass, circulating lipids and cardiovascular biomarkers (highly sensitive c-reactive protein (hs-CRP), N-terminal prohormone of brain natriuretic peptide (NT-proBNP), tumor necrosis factor-alpha (TNF-alpha), adiponectin and plasminogen activator inhibior-1 (PAI-1))
Changes in gut microbiota | baseline to 52 and 260 wks
  optional to the main protocol
Changes in subjective appetite | baseline to 52, 53, 260, and 261 wks
  visual analogue scale (VAS)
Number of participants with treatment-related adverse events (Safety and tolerability) | baseline to 52 and 260 wks
  as assessed by validated questionnaires
Change in Quality of life | Baseline to 52 and 260 wks
  Assessed by validated questionnaires (SF-36)
Evaluation of alcohol consumption | baseline to 52 and 260 wks
  By validated questionnaires
Evaluation of microalbuminuria | baseline to 52 to 260 wks
  Predicitve value of biomarkers for detection of microalbuminuria
Evaluation of blindedness of participants and investigators | baseline to 52 wks
  questionnaire and the end of the blinded trial
Changes in bonemarkers | baseline to 52 and 260 wks

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD, DMSc, Principal Investigator — University Hospital Gentofte; Signe Foghsgaard, MD, PhD, Principal Investigator — University Hospital Gentofte; Emilie Skytte Andersen, MD, PhD-student, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Clinical Metabolic Physiology, Steno Diabetes Center Copenhagen, Hellerup, Denmark

REFERENCES:
- [Background] Porte D Jr. Mechanisms for hyperglycemia in the metabolic syndrome. The key role of beta-cell dysfunction. Ann N Y Acad Sci. 1999 Nov 18;892:73-83. doi: 10.1111/j.1749-6632.1999.tb07786.x. PMID 10842653
- [Background] Vilsboll T, Holst JJ. Incretins, insulin secretion and Type 2 diabetes mellitus. Diabetologia. 2004 Mar;47(3):357-366. doi: 10.1007/s00125-004-1342-6. Epub 2004 Feb 13. PMID 14968296
- [Background] Vilsboll T. On the role of the incretin hormones GIP and GLP-1 in the pathogenesis of Type 2 diabetes mellitus. Dan Med Bull. 2004 Nov;51(4):364-70. No abstract available. PMID 16009062
- [Background] Holst JJ. The physiology of glucagon-like peptide 1. Physiol Rev. 2007 Oct;87(4):1409-39. doi: 10.1152/physrev.00034.2006. PMID 17928588
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Damm P, Vestergaard H, Kuhl C, Pedersen O. Impaired insulin-stimulated nonoxidative glucose metabolism in glucose-tolerant women with previous gestational diabetes. Am J Obstet Gynecol. 1996 Feb;174(2):722-9. doi: 10.1016/s0002-9378(96)70456-8. PMID 8623813
- [Background] Jensen DM, Molsted-Pedersen L, Beck-Nielsen H, Westergaard JG, Ovesen P, Damm P. Screening for gestational diabetes mellitus by a model based on risk indicators: a prospective study. Am J Obstet Gynecol. 2003 Nov;189(5):1383-8. doi: 10.1067/s0002-9378(03)00601-x. PMID 14634573
- [Background] Metzger BE, Coustan DR. Summary and recommendations of the Fourth International Workshop-Conference on Gestational Diabetes Mellitus. The Organizing Committee. Diabetes Care. 1998 Aug;21 Suppl 2:B161-7. No abstract available. PMID 9704245
- [Background] Lauenborg J, Hansen T, Jensen DM, Vestergaard H, Molsted-Pedersen L, Hornnes P, Locht H, Pedersen O, Damm P. Increasing incidence of diabetes after gestational diabetes: a long-term follow-up in a Danish population. Diabetes Care. 2004 May;27(5):1194-9. doi: 10.2337/diacare.27.5.1194. PMID 15111544
- [Background] Xiang AH, Kjos SL, Takayanagi M, Trigo E, Buchanan TA. Detailed physiological characterization of the development of type 2 diabetes in Hispanic women with prior gestational diabetes mellitus. Diabetes. 2010 Oct;59(10):2625-30. doi: 10.2337/db10-0521. Epub 2010 Aug 3. PMID 20682697
- [Background] Hanna FW, Peters JR. Screening for gestational diabetes; past, present and future. Diabet Med. 2002 May;19(5):351-8. doi: 10.1046/j.1464-5491.2002.00684.x. PMID 12027921
- [Background] Bian X, Gao P, Xiong X, Xu H, Qian M, Liu S. Risk factors for development of diabetes mellitus in women with a history of gestational diabetes mellitus. Chin Med J (Engl). 2000 Aug;113(8):759-62. PMID 11776065
- [Background] Gerich JE. The genetic basis of type 2 diabetes mellitus: impaired insulin secretion versus impaired insulin sensitivity. Endocr Rev. 1998 Aug;19(4):491-503. doi: 10.1210/edrv.19.4.0338. PMID 9715377
- [Background] Forbes S, Taylor-Robinson SD, Patel N, Allan P, Walker BR, Johnston DG. Increased prevalence of non-alcoholic fatty liver disease in European women with a history of gestational diabetes. Diabetologia. 2011 Mar;54(3):641-7. doi: 10.1007/s00125-010-2009-0. Epub 2010 Dec 12. PMID 21153530
- [Background] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Background] Astrup A, Carraro R, Finer N, Harper A, Kunesova M, Lean ME, Niskanen L, Rasmussen MF, Rissanen A, Rossner S, Savolainen MJ, Van Gaal L; NN8022-1807 Investigators. Safety, tolerability and sustained weight loss over 2 years with the once-daily human GLP-1 analog, liraglutide. Int J Obes (Lond). 2012 Jun;36(6):843-54. doi: 10.1038/ijo.2011.158. Epub 2011 Aug 16. PMID 21844879
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Flint A, Raben A, Astrup A, Holst JJ. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998 Feb 1;101(3):515-20. doi: 10.1172/JCI990. PMID 9449682
- [Derived] Foghsgaard S, Vedtofte L, Mathiesen ER, Svare JA, Gluud LL, Holst JJ, Damm P, Knop FK, Vilsboll T. The effect of a glucagon-like peptide-1 receptor agonist on glucose tolerance in women with previous gestational diabetes mellitus: protocol for an investigator-initiated, randomised, placebo-controlled, double-blinded, parallel intervention trial. BMJ Open. 2013 Oct 30;3(10):e003834. doi: 10.1136/bmjopen-2013-003834. PMID 24176797
- See also: Main website for the University Hospital Gentofte — http://gentoftehospital.dk